CLINICAL TRIAL: NCT04218851
Title: A Phase 2, Open-Label, Non-Comparative Clinical Trial to Study the Safety and Efficacy of Posaconazole (POS, MK-5592) in Pediatric Participants Aged 2 to Less Than 18 Years With Invasive Aspergillosis
Brief Title: Posaconazole (MK-5592) Intravenous and Oral in Children With Invasive Aspergillosis (IA) (MK-5592-104)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5592-104; MK-5592-104 (Other: MSD); 2019-002267-10 (EudraCT Number)
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Posaconazole (Experimental): On Day 1 participants receive 2 administrations of posaconazole (POS) 6 mg/kg body weight by intravenous (IV) infusion. On Days 2 through 7, participants receive POS 6 mg/kg body weight once daily by IV infusion. Beginning at Day 8 up to Day 84, participants may transition to receiving an oral formulation, or they may remain on the IV formulation.
  Interventions: Drug: Posaconazole IV; Drug: Posaconazole PFS; Drug: Posaconazole tablet

INTERVENTIONS:
Drug: Posaconazole IV — Posaconazole (POS) 6 mg/kg body weight by IV infusion
  Other Names: MK-5592; SCH 056592; Noxafil®
Drug: Posaconazole PFS — Dosing based on weight-band taken orally
  Other Names: MK-5592; SCH 056592; Noxafil®
Drug: Posaconazole tablet — POS tablet 300 mg taken orally
  Other Names: MK-5592; SCH 056592; Noxafil®

SUMMARY:
This study will evaluate the safety, efficacy, and pharmacokinetics of posaconazole (POS) intravenous (IV) and oral formulations in pediatric participants 2 to <18 years of age with invasive aspergillosis (IA).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of possible, probable, or proven IA per modified 2008/2020 European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG) disease definitions
* Has one or more of pre-defined risks as per modified 2008 EORTC/MSG disease definitions
* Has a central line (e.g., central venous catheter, peripherally-inserted central catheter) in place or planned to be in place prior to beginning IV study treatment.
* Has clinical symptoms consistent with an acute episode of IA, defined as duration of clinical syndrome of <30 days.
* Participants weigh at least 10 kg, and may be of any race/ethnicity.
* During the intervention period and for at least 30 days after the last dose of study treatment, males agree to be abstinent from heterosexual intercourse or use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause).
* Female is not pregnant or breastfeeding, and is not a woman of child bearing potential (WOCBP) or is a WOCBP using a highly effective contraceptive method. A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention.

Exclusion Criteria:

* Has chronic (≥30 days' duration) IA, relapsed/recurrent IA, or refractory IA that has not responded to prior antifungal treatment.
* Has cystic fibrosis, pulmonary sarcoidosis, aspergilloma, or allergic bronchopulmonary aspergillosis
* Has a known hypersensitivity or other serious adverse reaction to any azole antifungal therapy, or to any other ingredient of the study treatment used.
* Has any known history of torsade de pointes, unstable cardiac arrhythmia or proarrhythmic conditions, a history of recent myocardial infarction, congenital or acquired QT prolongation, or cardiomyopathy in the context of cardiac failure within 90 days of time of first dose of study treatment.
* Has known hereditary fructose intolerance.
* Has a known hereditary problem of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Is or has an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.
* Is on artificial ventilation at the time of first dose of study treatment.
* Has received any treatment prohibited by the protocol.
* Has enrolled previously in the current study and been discontinued.
* Is not expected, in the opinion of the investigator, to survive for at least 1 month after the initiation of study treatment.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (29):
- United States (4):
  - Children's Hospital of Orange County ( Site 1409), Orange, California
  - Rady Children's Hospital-San Diego ( Site 1401), San Diego, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago ( Site 1402), Chicago, Illinois
  - Washington University ( Site 1403), St Louis, Missouri
- Belgium (3):
  - UCL St Luc ( Site 1000), Brussels, Bruxelles-Capitale, Region de
  - UZ Gent ( Site 1002), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 1001), Leuven, Vlaams-Brabant
- Greece (3):
  - Athens Childrens Hospital Aglaia Kyriakou ( Site 1052), Athens, Attica
  - University General Hospital of Thessaloniki "AHEPA" ( Site 1053), Thessaloniki, Central Macedonia
  - General Hospital of Thessaloniki "Ippokrateio" ( Site 1050), Thessaloniki
- Hungary (3):
  - BAZ Megyei Korhaz. Klinikai Onkologia es Sugarterapias Centrum ( Site 1101), Miskolc, Borsod-Abauj Zemplen county
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet ( Site 1103), Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet ( Site 1102), Budapest
- Israel (4):
  - Rambam Medical Center ( Site 1125), Haifa
  - Hadassah Ein Karem Hebrew University Medical Center ( Site 1127), Jerusalem
  - Chaim Sheba Medical Center ( Site 1126), Ramat Gan
  - Sourasky Medical Center ( Site 1128), Tel Aviv
- Italy (2):
  - Ospedale Regina Margherita ( Site 1150), Torino
  - Azienda Ospedaliera Universitaria Integrata ( Site 1151), Verona
- Mexico (2):
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Infectologia ( Site 1204), Monterrey, Nuevo León
  - Instituto Nacional de Pediatria ( Site 1200), Mexico City
- Peru (2):
  - Instituto Nacional de Enfermedades Neoplásicas ( Site 1251), Lima
  - Hospital Nacional Edgardo Rebagliati Martins ( Site 1250), Lima
- Russia (4):
  - Almazov National Medical Research Centre ( Site 1284), Saint Petersburg, Leningradskaya Oblast'
  - Dmitry Rogachev National Research Center ( Site 1275), Moscow, Moscow
  - Institute of Invasive Mycosis ( Site 1282), Saint Petersburg, Sankt-Peterburg
  - Institute of Child Hematology and Transpl n.a.R.M.Gorbacheva ( Site 1281), Saint Petersburg, Sankt-Peterburg
- South Korea (2):
  - Seoul National University Hospital ( Site 1326), Seoul
  - The Catholic University of Korea. Seoul St. Mary s Hospital ( Site 1325), Seoul

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Kang HJ, Arrieta AC, Dhooge C, Kelemen A, Macias-Parra M, Aranda L, Dinikina YV, Kassis I, Cesaro S, Shepherd A, Shah AK, Mackey T, Waskin H, Johnson MG. Phase 2, open-label, noncomparative clinical trial evaluating safety and efficacy of posaconazole in pediatric patients with proven/probable invasive aspergillosis or possible invasive fungal disease. Antimicrob Agents Chemother. 2026 Jan 27:e0130525. doi: 10.1128/aac.01305-25. Online ahead of print. PMID 41589852
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Male or female participants with a diagnosis of possible, probable, or proven invasive aspergillosis (IA) aged 2 to <18 years were enrolled in this study.
Groups:
- Age Cohort 1 (2 -< 12 Years Old); Age Cohort 2 (12 -< 18 Years Old): On Day 1 participants receive 2 administrations of posaconazole (POS) 6 mg/kg body weight by intravenous (IV) infusion. On Days 2 through 7, participants receive POS 6 mg/kg body weight once daily by IV infusion. Beginning at Day 8 up to Day 84, participants may transition to receiving an oral formulation, or they may remain on the IV formulation.
Period: Overall Study
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old)
Started | 14 | 17
Completed | 13 | 14
Not Completed | 1 | 3
Not completed — Death | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old) | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (2.7) | 14.5 (1.7) | 11.1 (4.4)
Age, Customized [Number; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 14 | 0 | 14
  Adolescents (12-17 years) | 0 | 17 | 17
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 7 | 16 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 8 | 17
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience One or More Treatment-related Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Treatment-related AEs were determined by the investigator to be related to the drug. The 95% confidence interval (CI) was based on the exact binomial method by Clopper- Pearson.
Time Frame: Up to 14 days after treatment (up to Day 102)
Population: All enrolled participants who received at least 1 dose of study treatment, regardless of their IA classification.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old)
Number analyzed (Participants) | 14 | 17
Percentage of participants | 14.3 (1.8) [1.8 to 42.8] | 29.4 (10.3) [10.3 to 56.0]

2. Secondary Outcome: Percentage of Participants Who Have a Favorable Global Clinical Response Through Week 6
Description: A global clinical response is assessed by the investigator as favorable if the participant is alive and has a complete response (CR) or partial response (PR). CR is defined as survival within the prespecified period of observation, resolution of all attributable symptoms and signs of disease, resolution of radiological lesion(s), and documented clearance of infected sites that are accessible to repeated sampling. PR is defined as survival within the prespecified period of observation, improvement in attributable symptoms and signs of disease, improvement of radiological lesion(s), and evidence of clearance of infected sites that are accessible to repeated sampling.
Time Frame: Up to week 6
Population: Participants who have possible, probable, or proven IA; receive at least 1 dose of study treatment; have at least 1 post-allocation observation subsequent to at least 1 dose of study treatment; and have baseline data for those analyses that require baseline data.
Measure: Number; unit: Percentage of participants
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old)
Number analyzed (Participants) | 14 | 17
Percentage of participants
  Success, Complete Response | 42.9 | 17.6
  Success, Partial Response | 21.4 | 52.9

3. Secondary Outcome: Percentage of Participants Who Have a Favorable Global Clinical Response Through Week 12
Description: as for outcome 2
Time Frame: Up to Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old)
Number analyzed (Participants) | 14 | 17
Percentage of participants
  Success, Complete Response | 57.1 | 41.2
  Success, Partial Response | 21.4 | 35.3

4. Secondary Outcome: Percentage of Participants Who Have a Relapse of Invasive Aspergillosis (IA) at Any Point After Achieving Favorable Global Clinical Response
Description: In participants who achieved favorable global clinical response, relapse of IA is defined as the re-emergence of clinical, radiographic, or other relevant abnormalities indicating IA.
Time Frame: Up to 28 days post-treatment (up to Day 116)
Population: Participants who have possible, probable, or proven IA; receive at least 1 dose of study treatment; have at least 1 post-allocation observation subsequent to at least 1 dose of study treatment; have baseline data for those analyses that require baseline data; and who have achieved a favorable global clinical response at the end of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old)
Number analyzed (Participants) | 12 | 13
Percentage of participants | 0 | 0

5. Secondary Outcome: Average Plasma Concentration (Cavg) of POS by Age Cohorts
Description: Steady state Cavg was determined by population PK analysis of plasma concentrations obtained pre-dose up to Week 12 for each of Cohorts 1 and 2, as well as the pooled Cohorts 1 and 2. Some participants had 2 Cavg parameter values (1 for IV dosing, 1 for oral dosing).
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: All treated participants who had at least 1 postdose plasma concentration obtained after receiving at least 5 days of treatment. Per protocol PK results were analyzed for each age cohort, as well as the pooled age cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Units Other Than Participants: Cavg value
Groups:
- Age Cohort 1 (2 -< 12 Years Old); Age Cohort 2 (12 -< 18 Years Old); Age Cohorts 1 and 2 (2 -< 18 Years Old): On Day 1 participants receive 2 administrations of posaconazole (POS) 6 mg/kg body weight by intravenous (IV) infusion. On Days 2 through 7, participants receive POS 6 mg/kg body weight once daily by IV infusion. Beginning at Day 8 up to Day 84, participants may transition to receiving an oral (PFS or tablet) formulation, or they may remain on the IV formulation.
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old) | Age Cohorts 1 and 2 (2 -< 18 Years Old)
Number analyzed (Participants) | 13 | 15 | 28
Number analyzed (Cavg value) | 16 | 25 | 41
ng/mL | 2590 (50.8) | 2770 (55.4) | 2700 (53.0)

6. Secondary Outcome: Minimum Plasma Concentration (Cmin) of POS by Age Cohorts
Description: Steady state Cmin was determined by population PK analysis of plasma concentrations obtained pre-dose up to Week 12 for each of Cohorts 1 and 2, as well as the pooled Cohorts 1 and 2. Some participants had 2 Cmin parameter values (1 for IV dosing, 1 for oral dosing).
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Units Other Than Participants: Cmin value
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old) | Age Cohorts 1 and 2 (2 -< 18 Years Old)
Number analyzed (Participants) | 13 | 15 | 28
Number analyzed (Cmin value) | 16 | 25 | 41
ng/mL | 1610 (66.3) | 1920 (63.9) | 1790 (64.7)

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of POS by Age Cohorts
Description: Steady state Cmax was determined by population PK analysis of plasma concentrations obtained pre-dose up to Week 12 for each of Cohorts 1 and 2, as well as the pooled Cohorts 1 and 2. Some participants had 2 Cmax parameter values (1 for IV dosing, 1 for oral dosing).
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Units Other Than Participants: Cmax value
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old) | Age Cohorts 1 and 2 (2 -< 18 Years Old)
Number analyzed (Participants) | 13 | 15 | 28
Number analyzed (Cmax value) | 16 | 25 | 41
ng/mL | 3620 (48.5) | 3610 (53.7) | 3610 (51.0)

8. Secondary Outcome: Area Under the Concentration Time Curve Over the Dosing Interval (AUCtau) of POS by Age Cohorts
Description: Steady state AUCtau was determined by population PK analysis of plasma concentrations obtained pre-dose up to Week 12 for each of Cohorts 1 and 2, as well as the pooled Cohorts 1 and 2. Some participants had 2 AUCtau parameter values (1 for IV dosing, 1 for oral dosing).
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Units Other Than Participants: AUCtau value
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old) | Age Cohorts 1 and 2 (2 -< 18 Years Old)
Number analyzed (Participants) | 13 | 15 | 28
Number analyzed (AUCtau value) | 16 | 25 | 41
ng*h/mL | 62200 (50.8) | 66400 (55.4) | 64700 (53.0)

9. Secondary Outcome: Time to Reach Cmax (Tmax) of POS by Age Cohorts
Description: Steady state Tmax was determined by population PK analysis of plasma concentrations obtained pre-dose up to Week 12 for each of Cohorts 1 and 2, as well as the pooled Cohorts 1 and 2. Some participants had 2 Tmax parameter values (1 for IV dosing, 1 for oral dosing).
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: as for outcome 5
Measure: Median (Full Range); unit: hr.
Units Other Than Participants: Tmax value
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old) | Age Cohorts 1 and 2 (2 -< 18 Years Old)
Number analyzed (Participants) | 13 | 15 | 28
Number analyzed (Tmax value) | 16 | 25 | 41
hr. | 1.68 [1.25 to 7.10] | 1.63 [1.30 to 7.40] | 1.63 [1.25 to 7.40]

10. Secondary Outcome: Average Plasma Concentration (Cavg) of POS by Formulation
Description: Steady-state Cavg was determined by population PK analysis from plasma concentration obtained pre-dose up to Week 12 for each of the POS formulations: IV, PFS and tablet. Some participants may have received more than 1 formulation, and results were only reported when N > 2.
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: All treated participants who had at least 1 postdose plasma concentration obtained after receiving at least 5 days of treatment. Per protocol PK results were analyzed for each POS formulation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Age Cohort 1 (2 -< 12 Years Old): IV Formulation; Age Cohort 1 (2 -< 12 Years Old): PFS Formulation; Age Cohort 1 (2 -< 12 Years Old): Tablet Formulation; Age Cohort 2 (12 -< 18 Years Old): IV Formulation; Age Cohort 2 (12 -< 18 Years Old): PFS Formulation; Age Cohort 2 (12 -< 18 Years Old): Tablet Formulation: On Day 1 participants receive 2 administrations of posaconazole (POS) 6 mg/kg body weight by intravenous (IV) infusion. On Days 2 through 7, participants receive POS 6 mg/kg body weight once daily by IV infusion. Beginning at Day 8 up to Day 84, participants may transition to receiving an oral (PFS or tablet) formulation, or they may remain on the IV formulation.
Arm/Group | Age Cohort 1 (2 -< 12 Years Old): IV Formulation | Age Cohort 1 (2 -< 12 Years Old): PFS Formulation | Age Cohort 1 (2 -< 12 Years Old): Tablet Formulation | Age Cohort 2 (12 -< 18 Years Old): IV Formulation | Age Cohort 2 (12 -< 18 Years Old): PFS Formulation | Age Cohort 2 (12 -< 18 Years Old): Tablet Formulation
Number analyzed (Participants) | 10 | 6 | 1 | 13 | 2 | 10
ng/mL | 2900 (51.6) | 2070 (38.0) | NA (NA) — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 2860 (45.8) | NA (NA) — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 2500 (72.7)

11. Secondary Outcome: Minimum Plasma Concentration (Cmin) of POS by Formulation
Description: Steady-state Cmin was determined by population PK analysis from plasma concentration obtained pre-dose up to Week 12 for each of the POS formulations: IV, PFS and tablet. Some participants may have received more than 1 formulation, and results were only reported when N > 2.
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Age Cohort 1 (2 -< 12 Years Old): IV Formulation | Age Cohort 1 (2 -< 12 Years Old): PFS Formulation | Age Cohort 1 (2 -< 12 Years Old): Tablet Formulation | Age Cohort 2 (12 -< 18 Years Old): IV Formulation | Age Cohort 2 (12 -< 18 Years Old): PFS Formulation | Age Cohort 2 (12 -< 18 Years Old): Tablet Formulation
Number analyzed (Participants) | 10 | 6 | 1 | 13 | 2 | 10
ng/mL | 1680 (74.8) | 1410 (44.8) | NA (NA) — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 1820 (56.5) | NA (NA) — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 1910 (80.5)

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of POS by Formulation
Description: Steady-state Cmax was determined by population PK analysis from plasma concentration obtained pre-dose up to Week 12 for each of the POS formulations: IV, PFS and tablet. Some participants may have received more than 1 formulation, and results were only reported when N > 2.
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Age Cohort 1 (2 -< 12 Years Old): IV Formulation | Age Cohort 1 (2 -< 12 Years Old): PFS Formulation | Age Cohort 1 (2 -< 12 Years Old): Tablet Formulation | Age Cohort 2 (12 -< 18 Years Old): IV Formulation | Age Cohort 2 (12 -< 18 Years Old): PFS Formulation | Age Cohort 2 (12 -< 18 Years Old): Tablet Formulation
Number analyzed (Participants) | 10 | 6 | 1 | 13 | 2 | 10
ng/mL | 4530 (39.2) | 2510 (36.3) | NA (NA) — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 4180 (38.8) | NA (NA) — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 2880 (69.3)

13. Secondary Outcome: Area Under the Concentration Time Curve Over the Dosing Interval (AUCtau) of POS by Formulation
Description: Steady-state AUCtau was determined by population PK analysis from plasma concentration obtained pre-dose up to Week 12 for each of the POS formulations: IV, PFS and tablet. Some participants may have received more than 1 formulation, and results were only reported when N > 2.
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Age Cohort 1 (2 -< 12 Years Old): IV Formulation | Age Cohort 1 (2 -< 12 Years Old): PFS Formulation | Age Cohort 1 (2 -< 12 Years Old): Tablet Formulation | Age Cohort 2 (12 -< 18 Years Old): IV Formulation | Age Cohort 2 (12 -< 18 Years Old): PFS Formulation | Age Cohort 2 (12 -< 18 Years Old): Tablet Formulation
Number analyzed (Participants) | 10 | 6 | 1 | 13 | 2 | 10
ng*h/mL | 69600 (51.6) | 49700 (38.0) | NA (NA) — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 68600 (45.8) | NA (NA) — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 60100 (72.7)

14. Secondary Outcome: Time to Reach Cmax (Tmax) of POS by Formulation
Description: Steady-state Tmax was determined by population PK analysis from plasma concentration obtained pre-dose up to Week 12 for each of the POS formulations: IV, PFS and tablet. Some participants may have received more than 1 formulation, and results were only reported when N > 2.
Time Frame: Pre-dose, Day 1, Weeks 1, 2, 4, 6, 9 and 12
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Age Cohort 1 (2 -< 12 Years Old): IV Formulation | Age Cohort 1 (2 -< 12 Years Old): PFS Formulation | Age Cohort 1 (2 -< 12 Years Old): Tablet Formulation | Age Cohort 2 (12 -< 18 Years Old): IV Formulation | Age Cohort 2 (12 -< 18 Years Old): PFS Formulation | Age Cohort 2 (12 -< 18 Years Old): Tablet Formulation
Number analyzed (Participants) | 10 | 6 | 1 | 13 | 2 | 10
hr | 1.50 [1.25 to 1.77] | 7.00 [6.50 to 7.10] | NA [NA to NA] — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 1.50 [1.30 to 1.63] | NA [NA to NA] — NA = Per protocol, summary statistics were not calculated where N are 2 or less values. | 7.20 [6.90 to 7.40]

15. Secondary Outcome: Percentage of Participants With Different Categories of Palatability After First Day of Treatment With the POS PFS Formulation
Description: Palatability was categorized on the first day (Day 8) on PFS based on responses by participants to a palatability questionnaire. Per protocol participants were pooled into a single treatment group. Palatability categories for taste are as follows: Very good; Good; Very bad; Neither good nor bad.
Time Frame: First day of PFS treatment (Day 8)
Population: Participants who completed the palatability questionnaire. Per protocol participants were pooled into a single treatment group.
Measure: Number; unit: Percentage of participants
Groups:
- Pooled Participants (Ages 2 - < 18 Years Old): On Day 1 participants receive 2 administrations of POS 6 mg/kg body weight by IV infusion. On Days 2 through 7, participants receive POS 6 mg/kg body weight once daily by IV infusion. Beginning at Day 8 up to Day 84, participants may transition to receiving an oral formulation, or they may remain on the IV formulation.
Arm/Group | Pooled Participants (Ages 2 - < 18 Years Old)
Number analyzed (Participants) | 10
Percentage of participants
  Very good | 20
  Good | 40
  Very bad | 10
  Neither good nor bad | 30

16. Secondary Outcome: Percentage of Participants With Different Categories of Palatability After Last Day of Treatment With the POS PFS Formulation
Description: Palatability was categorized on the last day (Day 85) on PFS based on responses by participants to a palatability questionnaire. Per protocol participants were pooled into a single treatment group Palatability categories for taste are as follows: Very good; Good; Very bad; Neither good nor bad.
Time Frame: Last day of PFS treatment (Day 85)
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Participants (Ages 2 - < 18 Years Old)
Number analyzed (Participants) | 10
Percentage of participants
  Very good | 10
  Good | 40
  Very bad | 10
  Neither good nor bad | 40

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): from enrollment up to 14 days after treatment (up to Day 100), and included those reported beyond the final Day 114 study visit. Adverse events (AEs); from treatment up to 14 days after treatment (up to Day 102).
Description: ACM population analyzed was all enrolled participants. AE population analyzed was all enrolled participants who received at least 1 dose of study treatment, regardless of their IA classification.
Groups:
- Age Cohort 1 (2 -< 12 Years Old); Age Cohort 2 (12 -< 18 Years Old): On Day 1 participants receive 2 administrations of POS 6 mg/kg body weight by IV infusion. On Days 2 through 7, participants receive POS 6 mg/kg body weight once daily by IV infusion. Beginning at Day 8 up to Day 84, participants may transition to receiving an oral formulation, or they may remain on the IV formulation.
Arm/Group | Age Cohort 1 (2 -< 12 Years Old) | Age Cohort 2 (12 -< 18 Years Old)
All-Cause Mortality (participants affected / at risk) | 2/14 | 4/17
Serious Adverse Events (participants affected / at risk) | 4/14 | 8/17
Other Adverse Events (participants affected / at risk) | 12/14 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Cohort 1 (2 -< 12 Years Old) (N=14) | Age Cohort 2 (12 -< 18 Years Old) (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Administration site extravasation (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral sepsis (Infections and infestations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Leukaemic infiltration extramedullary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Cohort 1 (2 -< 12 Years Old) (N=14) | Age Cohort 2 (12 -< 18 Years Old) (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Aplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (2) | 0 (0)
Oculogyric crisis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (5)
Neutropenic colitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 7 (12)
Chills (General disorders) | 1 (2) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Infusion site thrombosis (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (14) | 6 (6)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus interstitial nephritis (Infections and infestations) | 0 (0) | 1 (1)
BK virus infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 2 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infectious disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Viraemia (Infections and infestations) | 0 (0) | 1 (1)
Viral haemorrhagic cystitis (Infections and infestations) | 0 (0) | 1 (1)
Viruria (Infections and infestations) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (7)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (5)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Kidney enlargement (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (5) | 5 (5)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT04218851/Prot_SAP_000.pdf